CLINICAL TRIAL: NCT00124566
Title: Three-Arm Randomized Phase II Clinical Study of Irofulven/Prednisone, Irofulven/Capecitabine/Prednisone or Mitoxantrone/Prednisone in Docetaxel-Pretreated Hormone-Refractory Prostate Cancer Patients
Brief Title: Study of Irofulven in Patients With Hormone-refractory Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Eisai Medical Services, Eisai Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IROF-018
Record Dates: First submitted 2005-07-26; First posted 2005-07-28 (Estimated); Last update posted 2016-01-18 (Estimated); Status verified 2016-01

CONDITIONS: Prostate Cancer
Keywords: Irofulven; Docetaxel; Taxotere
MeSH Terms: conditions — Prostatic Neoplasms | interventions — irofulven; Prednisone; Mitoxantrone; Capecitabine

ARMS (3):
- 1 (Experimental): Irofulven + prednisone
  Interventions: Drug: Irofulven; Drug: Prednisone
- 2 (Experimental): Irofulven + capecitabine + prednisone
  Interventions: Drug: Prednisone; Drug: Capecitabine; Drug: Irofulven
- 3 (Active Comparator): Mitoxantrone + prednisone
  Interventions: Drug: Prednisone; Drug: Mitoxantrone

INTERVENTIONS:
Drug: Irofulven — Subjects will receive irofulven in a 30 minute intravenous (IV) infusion at a dose of 0.45 mg/kg on Days 1 and 8 every 3 weeks.
  Arms: 1
Drug: Prednisone — Subjects will also receive oral prednisone at a dose of 10 mg per day in the morning.
Drug: Mitoxantrone — Subjects will receive mitoxantrone in an intravenous (IV) infusion (5 to 15 minutes) at a dose of 12 mg/m^2 per day, once every 3 weeks.
  Arms: 3
Drug: Capecitabine — Subjects will receive oral capecitabine at a dose of 1000 mg/m^2 twice daily for 15 days every 28 days.
  Arms: 2
Drug: Irofulven — Subjects will receive irofulven in a 30 minute intravenous (IV) infusion at a dose of 0.4 mg/kg on Days 1 and 15 every 4 weeks.
  Arms: 2

SUMMARY:
The purpose of this study is to assess the efficacy and safety of irofulven-based regimens compared to mitoxantrone plus prednisone in patients with hormone-refractory prostate cancer (HRPC) whose disease has progressed following Taxotere based regimens.

DETAILED DESCRIPTION:
For every five patients randomized, two will receive treatment number 1 (irofulven + prednisone), two patients will receive treatment number 2 (irofulven + capecitabine (Xeloda®) + prednisone), and one patient will receive treatment number 3 (mitoxantrone + prednisone). This is not a blinded study, so both the patient and doctor will know which treatment has been assigned.

ELIGIBILITY:
Inclusion Criteria:

To be included in the study, patients must meet the following criteria:

1. Cancer of the prostate confirmed by a biopsy sample.
2. 18 years of age or older.
3. Disease must have spread beyond the prostate as proven by chest x ray, abdominal and pelvic computed tomography (CT) scan, bone scan or clinical examination.
4. At least one prior hormonal treatment with documented disease progression during hormone therapy.
5. One previous line of chemotherapy that included Taxotere® (as monotherapy or in combination). This could be in addition to estramustine single agent therapy.
6. Disease progression during prior Taxotere-based therapy or within 3 months of discontinuing.
7. Recovered from any toxic effects of prior chemotherapy, radiotherapy and surgery.
8. Recovered from any toxic effects associated with other investigational drugs, if applicable.
9. Signed informed consent obtained prior to initiation of any study-specific procedures or treatment.

Exclusion Criteria:

Patients cannot participate in the study if any of the following apply:

1. Unable to use prednisone.
2. Prior treatment with irofulven, capecitabine (Xeloda), continuous/protracted infusion 5-FU (5-fluorouracil) (infusion duration greater than or equal to 24 hours), other fluoropyrimidines or mitoxantrone.
3. Ongoing treatment with a corticosteroid at a prednisone-equivalent dose > 10 mg/day.
4. More than 1 prior treatment with either 153Sm or 89Sr, or radioisotope treatment within 8 weeks prior to entering this study.
5. Initiation of treatment with bisphosphonate agents (e.g., pamidronate, etidronate) within 2 months of entering the study. Pre-existing treatment with bisphosphonate agents is to be continued during this study.
6. Treatment with warfarin and/or phenytoin within 14 days before entering this study or during the study period.

Please note: There are additional inclusion/exclusion criteria. The study center will determine if patients meet all of the criteria. If patients do not qualify for the trial, study personnel will explain the reasons. If patients do qualify, study personnel will explain the trial in detail and answer any questions. Patients can then decide if they wish to participate.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2004-06; Primary Completion 2006-01 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Time to progression: RECIST (Response Evaluation Criteria in Solid Tumors) criteria | Between randomization and study discontinuation or disease progression, whichever occurs later.
Time to progression: Prostate-specific antigen (PSA) evolution (Prostate-Specific Antigen Working Group Recommendations [PSAWGR criteria]). | Between randomization and study discontinuation or disease progression, whichever occurs later.

SECONDARY OUTCOMES:
Efficacy: Overall survival; objective response rate and PSA response rate according to RECIST and PSAWGR criteria, respectively. | Between randomization and death.
Determine safety profile of each treatment arm: incidence and severity of adverse events (AEs), serious AEs, and laboratory abnormalities. | Between randomization until a minimum of 30 days after last dose of study drug; treatment-related AEs will be followed until resolution.
Assess pain response in patients with significant pain at baseline using Tannock criteria and McGill-Melzack Pain Questionnaire. | Seven days prior to randomization and prior to each new cycle of study drug administration.
Quality of life (QOL) as measured by the Prostate Cancer Specific Quality of Life Instrument (PROSQOLI). | Between baseline and study drug discontinuation.

CONTACTS AND LOCATIONS:
Locations (50):
- United States (29):
  - Hot Springs, Arkansas
  - Jonesboro, Arkansas
  - Greenbrae, California
  - Colorado Springs, Colorado
  - Bonita Springs, Florida
  - Bradenton, Florida
  - Cape Coral, Florida
  - Fort Meyers, Florida
  - Naples, Florida
  - Port Charlotte, Florida
  - Sarasota, Florida
  - Venice, Florida
  - Atlanta, Georgia
  - Augusta, Georgia
  - Macon, Georgia
  - Marietta, Georgia
  - Chicago, Illinois
  - Minneapolis, Minnesota
  - Billings, Montana
  - Albany, New York
  - East Setauket, New York
  - Kettering, Ohio
  - Greenville, South Carolina
  - Nashville, Tennessee
  - Dallas, Texas
  - Fort Worth, Texas
  - Tyler, Texas
  - Spokane, Washington
  - Marshfield, Wisconsin
- Brazil (3):
  - Belo Horizonte
  - Porto Alegre
  - Rio de Janeiro
- Canada (5):
  - Calgary, Alberta
  - Vancouver, British Columbia
  - Winnipeg, Manitoba
  - London, Ontario
  - Montreal, Quebec
- Santiago, Chile
- Zagreb, Croatia
- France (5):
  - Avignon
  - Orléans
  - Paris
  - Saint-Brieuc
  - Saint-Grégoire
- Lima, Peru
- Romania (2):
  - Bucharest
  - Cluj-Napoca
- Russia (3):
  - Arkhangelsk
  - Chelyabinsk
  - Moscow